CLINICAL TRIAL: NCT02008695
Title: Youth and Adult Microfinance to Improve Resilience Outcomes in Democratic Republic of Congo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NA_00067820; R01HD071958 (NIH)
Record Dates: First submitted 2013-10-07; First posted 2013-12-11 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Mental Health Disorders
Keywords: Health; Youth; Microfinance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Youth microfinance only (Active Comparator): Youth receive loan
  Interventions: Behavioral: adult microfinance
- youth and adult micro finance (Active Comparator): youth and adult receive loan
  Interventions: Behavioral: Youth microfinance only
- adult microfinance (Active Comparator): adults receive loan
  Interventions: Behavioral: youth and adult micro finance

INTERVENTIONS:
Behavioral: adult microfinance — Female piglet provided to household member. Participants agrees to repay participants' "loan" by giving two piglets (one to repay the loan and one for the interest on the loan) to the association from the first litter of piglets (on average 6-12 piglets). These piglets are then given to other village member households
  Arms: Youth microfinance only
Behavioral: Youth microfinance only — One child (10-15 years) receive rabbits loan. The child is mentored by microfinance and community mentors. The child repays the loan to program and other children in the family and community are provided a loan from the repayment.
  Arms: youth and adult micro finance
Behavioral: youth and adult micro finance — One child and adult member of household receive animal loan. The child and adult are mentored and repayment of the loan to the program is provided and the repayment animal is provided to other members of the community
  Arms: adult microfinance

SUMMARY:
The investigators will test the effectiveness of a youth-led animal husbandry microfinance program, Rabbits for Resilience, combined with the adult microfinance, Pigs for Peace (PFP), program on youth, family and community resilience outcomes. The following aims will be completed over the five-year longitudinal, mixed-method, cluster randomized community trial:

Specific Aim 1: Determine the relative effectiveness of a youth-led microfinance combined with the adult microfinance on youth and family resilience outcomes (reduced mental health distress, increased economic stability, improved family functioning) compared to a youth-led microfinance only and adult microfinance only approaches.

* The investigators hypothesize that at six, twelve and 18-months post-baseline youth and adults in households in the youth-led and adult microfinance approach will report improved individual and family resilience outcomes compared to households in the youth-led microfinance only and adult microfinance only approaches.

Specific Aim 2: Determine the relative effectiveness of a youth-led microfinance combined with PFP microfinance on community resilience (e.g. social capital and participation in community groups by youth and adults) compared to youth-led microfinance only and adult microfinance only approaches.

* The investigators hypothesize that at 18-months post baseline in households in the youth-led and adult microfinance will report improved community resilience compared to households in the youth-led microfinance only and adult microfinance only approaches

Specific Aim 3: Determine if changes in youth resilience (caregiving ability, empathy and outlook for the future) mediate the relationship between youth engagement in microfinance and outcomes, as measured by reduced mental health distress, improved family functioning and improved social capital.

Specific Aim 4: Examine youth perspectives on resilience in the context of multiple adversities (war, poverty, loss of family, displacement, victimization). Youth participants (N=50, ages 10-15 years) will be invited (with parent/caregiver consent) to complete at baseline and 18 month post-baseline qualitative interview/group discussion to examine individual, family and community resilience and what that participants perceive as key to buffering the negative health and social consequences of prolonged conflict and other adversities.

DETAILED DESCRIPTION:
Congolese youth, families and communities have survived the 16 years of conflict and are now faced with significant challenges for rebuilding participants' futures. Developing, implementing and evaluating microfinance programs that combine youth and adults is an innovative strategy to assist households and community efforts by focusing on existing strengths. The study will advance knowledge for youth, families and communities impacted by armed conflicts in six critical areas:

* 1) increase the investigators' knowledge of youth and adult resilience (mental and physical health, family functioning, social capital) in context of multiple adversities;
* 2) measurement of resilience from a social ecological and longitudinal, mixed-method perspective;
* 3) expand investigators' understanding of resilience to develop prevention interventions for youth in early adolescence (ages 10-15 years), an important time to develop healthy transitions to young adulthood (ages 15-10 years);
* 4) test a youth-led microfinance program combined with an existing and successful adult microfinance program, Pigs For Peace (PFP), that is sustainable and appropriate to the context of a war-affected population;
* 5) detail resources and infrastructure needed for conducting research in challenging field settings with diverse cultures and languages as well as with limited resources, such as access to mental health professionals;
* 6) provide guidelines for the ethical conduct of research in settings where participants of diverse ages and backgrounds may have limited knowledge of human rights and ethical research concepts, such as informed consent and assent.

ELIGIBILITY:
Inclusion Criteria:

* girls/boys (ages 10-15 years) and women/men head of households (ages 16 years and older)
* Resident in participating 10 village in Walungu Territory in Democratic Republic of Congo

Exclusion Criteria:

* girls/boys under 10 years of age

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 988 (Actual)
Dates: Start 2012-08; Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Change in baseline Mental health distress at 18 months | Baseline to 18 months post baseline
  The outcome will be collected from multiple sources: 1) one randomly selected program eligible youth; and 2) one parent/caregiver in participating household

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Glass, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- PAIDEK, Congo, Bukavu, Republic of the Congo

REFERENCES:
- [Derived] Glass N, Remy MM, Mayo-Wilson LJ, Kohli A, Sommer M, Turner R, Perrin N. Comparative effectiveness of an economic empowerment program on adolescent economic assets, education and health in a humanitarian setting. BMC Public Health. 2020 Feb 4;20(1):170. doi: 10.1186/s12889-020-8219-6. PMID 32019539
- [Derived] Kohli A, Perrin NA, Remy MM, Alfred MB, Arsene KB, Nadine MB, Heri BJ, Clovis MM, Glass N. Adult and adolescent livestock productive asset transfer programmes to improve mental health, economic stability and family and community relationships in rural South Kivu Province, Democratic Republic of Congo: a protocol of a randomised controlled trial. BMJ Open. 2017 Mar 14;7(3):e013612. doi: 10.1136/bmjopen-2016-013612. PMID 28292764